CLINICAL TRIAL: NCT05385224
Title: A Clinical Study to Evaluate Effectiveness and Safety of the PillSense System in Detecting Blood in the Stomach for the Evaluation of Upper Gastrointestinal Bleeding (UGIB)
Brief Title: PillSense System for Detecting UGI Bleed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EnteraSense Limited (Industry)
Collaborators: Databean (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP-019-03
Record Dates: First submitted 2022-03-22; First posted 2022-05-23 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: UGI Bleed; Upper Gastrointestinal Bleeding; Upper Gastrointestinal Bleed
Keywords: EnteraSense; PillSense; UGI Bleed; UGIB; Upper Gastrointestinal Bleeding; Upper Gastrointestinal Bleed; Upper Gastrointestinal
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PillSense (Active) (Experimental): This is a single-arm, non-randomized study.
  Interventions: Diagnostic Test: PillSense

INTERVENTIONS:
Diagnostic Test: PillSense — The PillSense System is intended to detect the presence of blood in the stomach for the evaluation of upper gastrointestinal bleeding.

SUMMARY:
This is a prospective, non-randomized, open-label clinical investigation to evaluate feasibility, effectiveness and safety of the PillSense System, the transit of the PillSense Capsule through the GI tract, patient tolerability of the PillSense Capsule, and blood detection.

DETAILED DESCRIPTION:
Patient eligibility as set out in the inclusion/exclusion criteria for the clinical investigation will be reviewed prior to study enrollment. Prior to administering the PillSense Capsule, the PillSense Receiver will be paired with the PillSense Capsule. The PillSense Receiver collects and displays real-time information gathered by the PillSense Capsule. The PillSense Receiver interprets the data and displays a result message "Blood detected" or "No Blood detected". The overall investigation from the PillSense Capsule activation and ingestion until the result message is displayed takes less than 10 minutes. Esophagogastroduodenoscopy (EGD) should be completed immediately or up to 4 hours after PillSense Capsule administration in each patient that receives a "Blood detected" or "No blood detected" result to confirm the result achieved with the PillSense System. The endoscopy will be conducted according to the site's standard of care. Prior to discharge each patient will undergo an X-Ray examination to evaluate for PillSense Capsule presence. Following discharge, if there is no verifiable evidence that the PillSense Capsule passed through the gastrointestinal tract (GIT) (such as a photograph of stool with capsule in it or photograph of the capsule alone), the patient may undergo an X-Ray examination at Day 7 ± 5 days and, if necessary, at Day 14± 7 days to ascertain the passage status of the PillSense Capsule. If the PillSense Capsule did not pass through the GIT, it should be removed by an endoscopic method.

ELIGIBILITY:
Inclusion Criteria

* Age >=18 years
* Ability to provide informed consent
* Clinical suspicion of UGIB

Exclusion Criteria:

* Circulatory or hemodynamic instability
* Known GI tract stricture
* Using an implantable electrical device
* Difficulties in swallowing pills the size of the capsule
* History of: achalasia or known esophageal dysmotility; gastroparesis; severe constipation; Crohn's disease; bowel obstruction
* Currently taking medications intended for stimulation of GI motility
* Currently pregnant or breastfeeding, or intend to become pregnant during the investigation
* Suspected or previously diagnosed obstructing gastrointestinal tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Collins, Study Director — Technical Operations Director
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akiki K, Mahmoud T, Alqaisieh MH, Sayegh LN, Lescalleet KE, Abu Dayyeh BK, Wong Kee Song LM, Larson MV, Bruining DH, Coelho-Prabhu N, Buttar NS, Sedlack RE, Chandrasekhara V, Leggett CL, Law RJ, Rajan E, Gleeson FC, Alexander JA, Storm AC. A novel blood-sensing capsule for rapid detection of upper GI bleeding: a prospective clinical trial. Gastrointest Endosc. 2024 May;99(5):712-720. doi: 10.1016/j.gie.2023.11.051. Epub 2023 Dec 6. PMID 38065512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled between December 10, 2021 and August 18, 2022 at the Mayo Clinic, Rochester, MN.
Period: Overall Study
Arm/Group | PillSense (Active)
Started | 131
Modified Intent-to-Treat (Effectiveness Population) | 124
Safety Population | 126
Completed | 126
Not Completed | 5
Not completed — Unable to swallow capsule | 2
Not completed — Withdrawal by Subject | 2
Not completed — Did not meet study criteria | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | PillSense (Active)
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 122
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 117
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 126

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: To assess the sensitivity of the PillSense System in detecting the presence of blood in the stomach. The investigational device returns a result of either "Blood detected" or "No blood detected". Sensitivity = True Positives / (True Positives + False Negative). True positives were observations of bleed detected via PillSense capsule confirmed via esophagogastroduodenoscopy (EGD)]. False negatives were observation of bleed not detected via capsule but EGD confirmed bleed.
Time Frame: Day 1
Population: modified Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | PillSense (Active)
Number analyzed (Participants) | 28
Participants | 26

2. Primary Outcome: Specificity
Description: To evaluate the specificity of the PillSense System in detecting the presence of blood in the stomach. The investigational device returns a result of either "Blood detected" or "No blood detected". Specificity=True Negatives / (True Negatives + False Positive). True negatives were observations of no bleed detected via PillSense capsule confirmed via esophagogastroduodenoscopy (EGD)]. False positives were observation of bleed detected via capsule but EGD confirmed no bleed.
Time Frame: Day 1
Population: modified Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | PillSense (Active)
Number analyzed (Participants) | 96
Participants | 87

3. Secondary Outcome: NPV
Description: Negative predictive value (NPV) for the PillSense System in detecting the presence of blood in the stomach. The investigational device returns a result of either "Blood detected" or "No blood detected".
Time Frame: Day 1
Population: True Negatives + False Negatives
Measure: Count of Participants; unit: Participants
Arm/Group | PillSense (Active)
Number analyzed (Participants) | 89
Participants | 87

4. Secondary Outcome: Transit
Description: To evaluate the transit of the PillSense Capsule through the GI tract. Passage of the capsule will be monitored until capsule has passed from the body. If subject or study team is unable to determine capsule passage visually, a confirmation x-ray or other imaging will be used to determine if the capsule is still present in the body.
Time Frame: Day 1 through Day 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PillSense (Active)
Number analyzed (Participants) | 126
days | 3.6 (2.35)

5. Secondary Outcome: PPV
Description: Positive predictive value (PPV) for the PillSense System in detecting the presence of blood in the stomach. The investigational device returns a result of either "Blood detected" or "No blood detected".
Time Frame: Day 1
Population: True Positives + False Positives
Measure: Count of Participants; unit: Participants
Arm/Group | PillSense (Active)
Number analyzed (Participants) | 35
Participants | 26

ADVERSE EVENTS:
Time Frame: From Time of PillSense Administration through Follow-up Visit 3 (Up to 21 days).
Description: Treatment emergent adverse events defined as an adverse event that began or worsened during or after PillSense Capsule administration.
Arm/Group | PillSense (Active)
All-Cause Mortality (participants affected / at risk) | 0/126
Serious Adverse Events (participants affected / at risk) | 15/126
Other Adverse Events (participants affected / at risk) | 9/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PillSense (Active) (N=126)
Suicidal Ideations (Psychiatric disorders) | 1 (1)
Alchohol withdrawal seizure (Social circumstances) | 2 (2)
Abdominal Distention / Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Bleeding (Gastrointestinal disorders) | 5 (5)
Altered Mental Status (Nervous system disorders) | 1 (1)
Chest Pain with SOB (Cardiac disorders) | 1 (1)
Acute Limb Ischemia (Vascular disorders) | 1 (1)
Amyloidosis and Multiple Myeloma (Blood and lymphatic system disorders) | 1 (1)
Hemobilia (Hepatobiliary disorders) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Failure to extubate (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PillSense (Active) (N=126)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Lethargy (General disorders) | 1 (1)
Lumbar Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Epistasix (Ear and labyrinth disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT05385224/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT05385224/SAP_001.pdf